CLINICAL TRIAL: NCT06361121
Title: Analgesic Efficacy of Mid-point Transverse Process to Pleura Block Compared With Thoracic Paravertebral Block in Adult Patients Undergoing Posterolateral Thoracotomy Incisions: A Randomized Controlled Study
Brief Title: Mid-point Transverse Process to Pleura Block Versus Thoracic Paravertebral Block in Posterolateral Thoracotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D361
Record Dates: First submitted 2024-03-27; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Bronchiectasis; Lung Neoplasm; Emphysematous Bleb of Lung
Keywords: Mid-point Transverse Process to Pleura Block; Posterolateral Thoracotomy Incisions
MeSH Terms: conditions — Bronchiectasis; Lung Neoplasms | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients will be randomized into two groups: MTP block group and TPV block group in a 1:1 ratio using a computer-generated random table. The patient's assigned group information will be elicited from a sealed opaque envelope by the anesthesiologist who will perform the US-guided MTP and TPV block and will not be involved in further data collection or patient care. The patients and both the surgical and anesthesia teams, who are responsible for patient care and data collection are blinded from the group assignments
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mid-point transverse process to pleura (MTP) block (Active Comparator): In MTP block group, A 22G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the 2 transverse processes and advanced till it reaches the mid-point between the transverse process and pleura. After negative aspiration of blood or air, a total volume of 20 ml of bupivacaine 0.25% ( not exceeding a maximum dose of 2 mg/kg) will be injected superficial to the SCTL
  Interventions: Procedure: mid-point transverse process to pleura (MTP) block
- Thoracic Paravertebral (TPV) Block (Active Comparator): In the TPV block group , the transverse process and the pleura will be identified and the needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space. After negative aspiration of blood or air a total volume of 20 ml of bupivacaine 0.25% will be injected displacing the pleura downwards
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: mid-point transverse process to pleura (MTP) block — the T1-T12 thoracic spinal levels will be sonographically identified using a high frequency linear US probe (HFL_50, 15_6MHz). Then the probe will be placed vertically and nearly 3 cm lateral to the spinous process at the thoracic level T4/T5. The paraspinal muscles (erector spinae, trapezius, rhomboid), transverse processes , superior costo-transverse ligament (SCTL) and parietal pleura will be all identified under parasagittal scanning.
  In MTP block group, A 22G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the 2 transverse processes and advanced till it reaches the mid-point between the transverse process and pleura. After negative aspiration of blood or air, a total volume of 20 ml of bupivacaine 0.25% ( not exceeding a maximum dose of 2 mg/kg) will be injected superficial to the SCTL.
  Arms: mid-point transverse process to pleura (MTP) block
Procedure: Thoracic Paravertebral Block — In the TPV block group , the transverse process and the pleura will be identified and the needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space. After negative aspiration of blood or air a total volume of 20 ml of bupivacaine 0.25% will be injected displacing the pleura downwards
  Arms: Thoracic Paravertebral (TPV) Block

SUMMARY:
The ultrasound guided Thoracic paravertebral (TPV) block in the context of posterolateral thoracotomy offers targeted pain relief by anesthetizing the spinal nerves as they emerge from the intervertebral foramina, producing ipsilateral somatosensory, visceral and sympathetic nerve blockade. TPV block involves the injection of local anesthetic (LA) into the wedge-shaped paravertebral space deep to the superior costotransverse ligament (SCTL)

Costach et al introduced the mid-point transverse process to pleura block (MTP) as a modification of conventional paravertebral block by placing the LA posterior to the (SCTL) under ultrasound guidence achieving an effective block without the necessity to approach the pleura and the attendant risks.

In recent studies ,the ultrasound guided MTP block provided an effective analgesia in various surgical procedures including mastectomy , video-assisted thoracic surgeries and cardiac surgeries.

In our study we hypothesized that the mid-point transverse process to pleura (MTP) block can provide an effective analgesia comparable with thoracic paravertebral (TPV) block in adult patients undergoing posterolateral thoracotomy incisions.

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board. Patients who are scheduled for elective thoracic surgeries via posterolateral thoracotomy incision and fulfilling the inclusion criteria in Fayoum university hospital starting from March 2024 will be enrolled in this randomized controlled study until fulfilling sample size. A detailed informed consent will be signed by the eligible participants before recruitment.

The patients will be randomized into two groups: MTP block group and TPV block group in a 1:1 ratio using a computer-generated random table. The patient's assigned group information will be elicited from a sealed opaque envelope by the anesthesiologist who will perform the US-guided MTP and TPV block and will not be involved in further data collection or patient care. The patients and both the surgical and anesthesia teams, who are responsible for patient care and data collection are blinded from the group assignments.

In this study, no premedication will be given to the patients before the operation. All patients will be monitored using electrocardiography, pulse-oximetry, capnography. An arterial line will be inserted using a 20 G cannula either right or left radial artery for invasive blood pressure monitoring in the operating room.

After pre-oxygenation, general anesthesia will be induced with intravenous propofol (2 mg/kg) and fentanyl (1 μg/kg). After muscle relaxation with atracurium (0.5mg/kg), tracheal intubation will be performed by a cuffed endotracheal tube (7-7.5) size and mechanical ventilation will be applied while maintaining the end-tidal CO2 between 30 and 35 mmHg. Maintenance of anesthesia will be made using inhalational anesthesia (isoflurane) and IV atracurium according to the patients' requirements. The anesthesia will be maintained with isoflurane starting at one MAC and will be adjusted to obtain an adequate level of anesthesia by titrating the concentration according to the BIS monitoring (BIS Complete Monitoring System P/N 185-0151 Covidien IIc, 15 Hampshire Street, Mansfield, MA 02048 USA) to keep the BIS value between 40 and 60.

After induction , the patient will be placed in the lateral decubitus position. The same anesthesiologist will perform the block.

In both groups, the T1-T12 thoracic spinal levels will be sonographically identified using a high frequency linear US probe (HFL_50, 15_6MHz). Then the probe will be placed vertically and nearly 3 cm lateral to the spinous process at the thoracic level T4/T5. The paraspinal muscles (erector spinae, trapezius, rhomboid), transverse processes , superior costo-transverse ligament (SCTL) and parietal pleura will be all identified under parasagittal scanning.

In MTP block group, A 22G, 50mm block needle (SONOTAP,Pajunk, -Geisingen,Germany) will be inserted in the cranial to caudal direction via an in-plane approach between the 2 transverse processes and advanced till it reaches the mid-point between the transverse process and pleura. After negative aspiration of blood or air, a total volume of 20 ml of bupivacaine 0.25% ( not exceeding a maximum dose of 2 mg/kg) will be injected superficial to the SCTL.

In the TPV block group , the transverse process and the pleura will be identified and the needle will be inserted in the cranial to caudal direction till it pierces the SCTL and reaches the paravertebral space. After negative aspiration of blood or air a total volume of 20 ml of bupivacaine 0.25% will be injected displacing the pleura downwards.

After 15 min , an incision will be made to perform the surgical procedure. . Continuous hemodynamic monitoring of blood pressure and heart rate will be done . If the systolic blood pressure decreased to a 20% below the baseline or less than 90 mmHg, 5 mg of ephedrine will be injected IV. Moreover, if the heart rate reduced to a 50 bpm or less, 0.5 mg of atropine will be injected IV.

At the end of the surgery, isoflurane will be discontinued and the muscle relaxant will be antagonized with neostigmine (0.04-0.08 mg/kg) and atropine (0.01 mg/kg) and will be extubated when the patient meets the following criteria: awake or arousable, hemodynamically stable, no ongoing active bleeding, warm extremities, no electrolyte abnormalities, and a satisfactory arterial blood gas , after the return of spontaneous respiration.

After admission to the Post-Anesthesia Care Unit (PACU) at the end of surgery, all patients will receive IV fentanyl via patient controlled analgesia (PCA) with concentration 10 μg/ml , with bolus 15 μg and lockout interval 10 minutes and maximum dose of 90 μg/hr with no background dose for 24 hours. Paracetamol 1 gm IV will be given every 8 hours.. The patient's pain will be evaluated using a Visual Analog Scale (VAS) both during rest and with cough (0: no pain, 10: worst pain ever) at time intervals: 30 minutes, 1 hour, 3 hours, 6 hours, 12 hours, and 24h postoperative. The total 24 h. fentanyl consumption will be calculated based on the volume remaining in the PCA after 24h based on the following formula : Total fentanyl consumption = (total volume - remaining volume )x 10

ELIGIBILITY:
Inclusion Criteria:

* Patients Scheduled for elective thoracic surgery for pneumectomy, lobectomy, bullectomy or pleural decortication via posterolateral thoracotomy incision.
* American Society of Anesthesiologists (ASA) physical status I-III patients

Exclusion Criteria:

* Patient refusal.
* Significant renal, hepatic and cardiovascular diseases.
* History of allergy to one of the study drugs.
* Any contraindication to regional anesthesia such as local infection or bleeding disorders.
* Chronic opioid use, history of chronic pain and cognitive disorders.
* Emergent or re-do surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The total postoperative fentanyl consumption | in the first 24 hours
  The total 24 h. fentanyl consumption will be calculated based on the volume remaining in the PCA after 24h based on the following formula : Total fentanyl consumption = (total volume - remaining volume )x 10 .

SECONDARY OUTCOMES:
Demographic data | 24 hours before operation
  :age, sex, body mass index, type of surgery and comorbidities
visual analogue scale score both during rest and with cough | from 30 minutes up to 24 hours postoperative
  (score 0 =no pain and 10 =worst pain ever) in the two groups of the study
intra operative fentanyl consumption | from induction of anesthesia to extubation
  Dose of administered fentanyl in micrograms
Duration of surgery | from induction of anesthesia to extubation
  Duration of surgery in minutes
Blood pressure | from induction of anesthesia up to 24 hours post operative
  measured blood pressure intraoperatively every 30 minutes and postoperatively every 6 hours
Heart rate | from induction of anesthesia up to 24 hours post operative
  Readings of heart rate intra operatively every 30 minutes and postoperatively every 6 hours
Oxygen saturation | from induction of anesthesia up to 24 hours post operative
  Readings of oxygen saturation intra operatively every 30 minutes and postoperatively every 6 hours
complications related to the block | from induction of anesthesia up to 24 hours post operatively
  Number of patients who developed hypotension (systolic blood pressure decreased to a 20% below the baseline or less than 90 mmHg) , Number of patients who developed bradycardia (heart rate reduced to a 50 bpm or less) , Incidence of pleural puncture or vascular puncture or local anesthesia systemic toxicity.
complications related to IV opioids | assessed up to 24 hours postoperatively
  Number of Participants with nausea and vomiting (0 = no symptoms, 1 = only nausea, 2 = nausea and vomiting), respiratory depression (respiratory rate less than 10), sedation (0 = awake and alert, 1 = quietly awake, 2 = asleep but easily arousable, 3 = deep sleep, responding to painful stimulus).
Hospital length of stay in days | the time elapsed from day 0; the operative day; to the time of discharge up to 30 days
  Days spent in hospital from operative day to day of discharge
Participant satisfaction | from the operative day; to the time of discharge up to 30 days
  will be assessed on a 4-point scale (1: excellent, 2: good 3: fair, 4: poor).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Fayoum University Hospital
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costache I, de Neumann L, Ramnanan CJ, Goodwin SL, Pawa A, Abdallah FW, McCartney CJL. The mid-point transverse process to pleura (MTP) block: a new end-point for thoracic paravertebral block. Anaesthesia. 2017 Oct;72(10):1230-1236. doi: 10.1111/anae.14004. Epub 2017 Aug 1. PMID 28762464
- [Background] Chin KJ, Versyck B, Pawa A. Ultrasound-guided fascial plane blocks of the chest wall: a state-of-the-art review. Anaesthesia. 2021 Jan;76 Suppl 1:110-126. doi: 10.1111/anae.15276. PMID 33426660
- [Background] Bhoi D, Narasimhan P, Nethaji R, Talawar P. Ultrasound-Guided Midpoint Transverse Process to Pleura Block in Breast Cancer Surgery: A Case Report. A A Pract. 2019 Feb 1;12(3):73-76. doi: 10.1213/XAA.0000000000000850. PMID 30085935
- [Background] Kahramanlar AA, Aksoy M, Ince I, Dostbil A, Karadeniz E. The Comparison of Postoperative Analgesic Efficacy of Ultrasound-Guided Paravertebral Block and Mid-Point Transverse Process Pleura Block in Mastectomy Surgeries: A Randomized Study. J Invest Surg. 2022 Sep;35(9):1694-1699. doi: 10.1080/08941939.2022.2098544. Epub 2022 Jul 17. PMID 35848451